CLINICAL TRIAL: NCT05659368
Title: Towards a Personalized Precision Medicine in Rare Disease: Tirzepatide (a Dual Glucose-dependent Insulinotropic Polypeptide and Glucagon-like Peptide-1 Receptor Agonist) Monotherapy in Patients With Wolfram Syndrome Type 1
Brief Title: Tirzepatide Monotherapy in Patients With Wolfram Syndrome Type 1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Lorenzo Piemonti, Principal Investigator, Ospedale San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Wolfram Tirzepatide; 2022-003853-70 (EudraCT Number); PNRR-MR1-2022-12375914 (Other Grant/Funding Number: National Recovery and Resilience Plan)
Record Dates: First submitted 2022-12-05; First posted 2022-12-21 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Wolfram Syndrome
Keywords: wolfram syndrome; diabetes; tirzepatide; insulin secretion
MeSH Terms: conditions — Wolfram Syndrome; Diabetes Mellitus | interventions — Tirzepatide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional group (Experimental): Tirzepatide will be injected subcutaneously once-per-week, in the abdomen, thigh or upper arm. To improve gastro-intestinal tolerability, the starting dose will be 5 mg (2.5mg for prepubertal children) and will be increased to a maximum of 15 mg (or highest tolerated dose).
  Interventions: Drug: Tirzepatide

INTERVENTIONS:
Drug: Tirzepatide — tirzepatide once weekly

SUMMARY:
Wolfram syndrome (WFS:OMIM 222300) is a group of inherited disorders that usually appear in childhood and cause diabetes, optic atrophy leading to loss of vision, deafness and often diabetes insipidus. Wolfram syndrome affected no more than 0.2 in 10,000 people in the European Union. There is no cure and no treatment that will arrest or delay the progress of the disease.

The gene responsible for WS1 is WFS1, it encodes for wolframin, a transmembrane glycoprotein involved in the regulation of the unfolded protein response. Recently, drug repurposing has been hypothesized from others and us as being useful for WS1 therapy. More specifically, GLP-1 receptor agonists were suggested as a promising class of anti- diabetic drugs having the potential to delay or even reverse disease progression based on their ability to reduce elevated ER stress in vitro and in vivo.

The objective of this project is to create a model of precision-medicine oriented Rare Diabetes Clinic, which will be specifically dedicated to the treatment and follow-up of complex patients with Wolfram Syndrome. A team of clinicians and researchers specialized in diabetes and/or optic neuropathy and with experience in the subset of monogenic forms will make available a cohort of subjects with Wolfram Syndrome prospectively followed in an interventional protocol on the use of tirzepatide (a dual glucose-dependent insulinotropic polypeptide and glucagon-like peptide-1 receptor agonist). It will be a prospective phase 2, non-randomized, single group assignment, intervention trial to determine the efficacy of tirzepatide (GIP/GLP-1 receptor agonist) in increasing endogenous insulin production and correcting glycemic lability in patients with Wolfram syndrome type 1 (WS1).

The expected outcomes of this study are 1) to provide a therapeutic option for a devastating orphan disease; 2) to confirm the efficacy of a repurposed drug able to reduce elevated endoplasmic reticulum (ER) stress in a disease that represents a model of ER disease; 3) to confirm the efficacy of the disease modeling based on iPSC to predict the response to treatment; 4) to develop a disease-specific multidisciplinary follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. A definitive diagnosis of Wolfram syndrome, as determined by the following:

   1. Documented diabetes mellitus diagnosed under 16 completed years according to WHO or ADA criteria AND
   2. Documented functionally relevant recessive mutations on both alleles of the WFS1 gene or dominant mutation on one allele of the WFS1 gene based on historical test results (if available) or from a qualified laboratory at screening;
2. Aged 5 years or older;
3. The patient, patient's parent(s), or legally authorized guardian(s) must have voluntarily signed an Institutional Review Board/Independent Ethics Committee-approved informed consent form after all relevant aspects of the study have been explained and discussed with the patient. The guardians' consent and patient's assent, as relevant, must be obtained;
4. Females of child bearing potential will only be included after a negative highly sensitive urine pregnancy test. If sexually active, they must agree to use a highly effective contraception measure;
5. Patient willing to wear a continuous glucose monitor.

Exclusion Criteria:

1. Clinically significant non-Wolfram related CNS involvement which is judged by the Investigator to be likely to interfere with the accurate administration and interpretation of protocol assessments;
2. A history of pancreatitis;
3. Pre-existing thyroid disease;
4. A personal or family history of medullary thyroid carcinoma;
5. Multiple Endocrine Neoplasia syndrome type 2;
6. Active liver or renal disease, personal or family history of liver/kidney dysfunction related to known genetic disorders;
7. Treatment with any investigational drug within the 30 days prior to Trial entry;
8. Current therapy with of GLP-1 agonist or DDP-4 inhibitor or a known hypersensitivity to GLP-1 agonist;
9. Any other acute or chronic medical, psychiatric, social situation or laboratory result that, based on investigator's judgment, would jeopardize patient safety during trial participation, cause inability to comply with the protocol, or affect the Trial outcome;
10. Breastfeeding;
11. Pre-existing ocular disease (corneal or lens diseases and any other retinal or optic nerve non-Wolfram related diseases).

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
changing in endogenous insulin production | [Time Frame: month 6±1, month 12±1]
  C-peptide response in the Mixed Meal Tolerance Test (MMTT; change from baseline C-peptide response)
changing in insulin production | [Time Frame: month 6±1, month 12±1]
  mean change from baseline in stimulated 2 hour plasma C-peptide AUC (from MMTT) maximum stimulated plasma C-peptide: the highest value at any time point during the MMTT

SECONDARY OUTCOMES:
glucose variability | [Time Frame: month 6±1, month 12±1]
  change from baseline in average glucose (measured by continuous glucose monitoring)
glycemic variability | [Time Frame: month 6±1, month 12±1]
  change from baseline in coefficient of glucose variation (measured by continuous glucose monitoring)
change in time in range | [Time Frame: month 6±1, month 12±1]
  change from baseline in time in range (measured by continuous glucose monitoring)
change in insulin requirements | [Time Frame: month 3±1, month 6±1, month 12±1]
  change from baseline in mean daily insulin use over the 3 days preceeding the study visits. The mean daily insulin use value will be calculated, in units of U/kg/day, as the mean of the values of amount of insulin used per day on each of the last three consecutive days preceeding each study visits.
change in HbA1c | [Time Frame: month 3±1, month 6±1, month 12±1]
  change from baseline in HbA1c

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Piemonti, MD, Principal Investigator — Ospedale San Raffaele
Locations (1):
- IRCCS San Raffaele Scientific Institute, Milan, Italy